CLINICAL TRIAL: NCT04806685
Title: Diabetes Education and A1c Study
Acronym: DEA1c
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Blue Cross Blue Shield Foundation of Michigan (Unknown)
Responsible Party: Principal Investigator, Robin Tucker, Assistant Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00005457
Record Dates: First submitted 2021-03-15; First posted 2021-03-19 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Diabetes Mellitus, Type 2; Sleep
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Diet therapy plus sleep education
  Interventions: Behavioral: Sleep education
- Control (Other): Diet therapy
  Interventions: Behavioral: Diet only

INTERVENTIONS:
Behavioral: Sleep education — Medical nutrition therapy plus behavior-based sleep education intervention
  Arms: Intervention
Behavioral: Diet only — No sleep education
  Arms: Control

SUMMARY:
Sleep problems are associated with poor blood glucose control, but current diabetes self-management programs do not include sleep education. This study will randomize participants into two groups: one that receives sleep education and one that does not. The researchers expect both groups to experience reductions in blood glucose. The researchers hypothesize that individuals who receive sleep education as part of their diabetes self-management training will experience greater improvements in blood glucose control, as measured by hemoglobin A1c, compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a diagnosis of type 2 diabetes who are patients at the Michigan State University (MSU) Endocrinology clinic,
* a diagnosis of overweight or obesity (Body Mass Index greater than or equal to 25.0 kg/m2),
* the most recent hemoglobin A1c value greater than or equal to 7.5%, and
* the ability to attend online program sessions.

Exclusion Criteria:

* significant psychiatric disorders,
* advanced medical conditions that require alterations to the MNT for DM2, e.g., advanced chronic kidney disease, and
* an inability to follow recommendations due to cognitive deficits.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c | 12 weeks
  Lab value

SECONDARY OUTCOMES:
Body mass index | 12 weeks
  Calculated from height and weight
Sleep duration | 12 weeks
  FitBit outcomes data
Sleep quality | 12 weeks
  Pittsburgh Sleep Quality Index
Diabetes self-care | 12 weeks
  Diabetes Self-Management Questionnaire
Epworth Sleepiness Scale | 12 weeks
  Validated survey measuring excessive daytime sleepiness
Insomnia Severity Index | 12 weeks
  Validated survey measuring insomnia symptoms

CONTACTS AND LOCATIONS:
Locations (1):
- Michigan State University, East Lansing, Michigan, United States